CLINICAL TRIAL: NCT02647190
Title: A Phase I Study to Determine the Safety and Pharmacokinetics of Intravenous Erwinia Chrysanthemi Asparaginase in Patients With Newly Diagnosed Philadelphia Chromosome Negative Acute Lymphoblastic Leukemia Aged 60 Years or Older
Brief Title: Intravenous Erwinia Chrysanthemi Asparaginase in Patients With Newly Diagnosed Philadelphia Chromosome Negative Acute Lymphoblastic Leukemia Aged 60 Years or Older
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-107
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Newly Diagnosed Philadelphia Chromosome Negative; Aged 60 Years or Older
Keywords: Erwinia Chrysanthemi Asparaginase; 15-107
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant

ARMS (1):
- Erwinia Chrysanthemi asparaginase (Experimental): This is a phase I trial designed to assess the safety of IV Erwinia Chrysanthemi asparaginase during initial induction in patients aged 60 years or older with newly diagnosed Ph-negative ALL. A total of 12 patients will be accrued to the study.
  Interventions: Drug: Erwinia Chrysanthemi asparaginase

INTERVENTIONS:
Drug: Erwinia Chrysanthemi asparaginase

SUMMARY:
The purpose of this study is to test the safety of Erwinia Chrysanthemi asparaginase when used alone and together with chemotherapy and find out what effects, if any, it has on people.

DETAILED DESCRIPTION:
The study consists of three treatment phases.

1. Steroid prophase (days -3 to -1):

   To prevent rapid leukemia progression and reduce tumor load, patients will receive either prednisone 60mg/m2 oral daily or equivalent corticosteroid daily for 3 days.
2. Asparaginase phase (days 1 - 14):

   Patients will receive Erwinia asparaginase 25,000 IU/m2 IV three times a week on a Monday, Wednesday, Friday (MWF) schedule for 2 weeks. Patients are permitted to begin Erwinia asparaginase on Monday, Wednesday, or Friday, so that their schedules are defined as MWF, WFM, or FMW. For rapid progression of disease (defined by rising WBC >30K with > 50% peripheral blasts), prednisone 60mg/m2 oral daily or equivalent corticosteroid daily may be added.

   Bone marrow aspirate and/or biopsy will be performed on days 13-15 of the asparaginase treatment for early disease response assessment.
3. Chemotherapy phase (days 15 - 42):

   * Cyclophosphamide 650 mg/m2 IV on day 15
   * Vincristine 1.4 mg/m2 (max 2mg) IV on days 15, 22, 29, and 36
   * Prednisone 60mg/m2 (or equivalent corticosteroid) oral daily for 28 days on days 15 - 42
   * Erwinia asparaginase 25,000 IU/m2 IV three times a week on a MWF schedule for 2 weeks on days 29 - 42 (after a two week interval without Erwinia asparaginase administered on days 1 - 14) Upon cell count recovery, a bone marrow aspirate and/or biopsy will be performed to assess the disease response. Subsequent treatments following the bone marrow evaluation will be left up to the discretion of the treating physicians. If the first 6 patients have no response or progress during the 2 weeks of asparaginase phase of treatment with or without steroid, the next 6 patients will start directly with the chemotherapy phase (days 15-42) of treatment consisting of cyclophosphamide, vincristine, and prednisone with Erwinia asparaginase.

CNS prophylaxis:

* IT methotrexate 12mg (flat dose) between days 15 - 22
* IT methotrexate 12mg (flat dose) between days 22- 29
* There will be a minimal interval between doses of 7 days

ELIGIBILITY:
Inclusion Criteria:

* Ages 60 years or older
* Previously untreated Philadelphia chromosome negative acute lymphoblastic leukemia
* No prior treatment for ALL, except steroids or hydroxyurea (stopped within 24 hour before start of protocol treatment)
* Serum creatinine ≤ 2 x upper limit of normal (ULN)
* Adequate liver function, including total bilirubin ≤ 1.5 x ULN unless the patient has documented Gilbert syndrome, and aspartate and alanine aminotransferase (AST and ALT) ≤ 5 x ULN. If organ function abnormalities are considered due to leukemic infiltration, total bilirubin must be ≤ 2 x ULN.
* ECOG performance status ≤3
* Male and female patients of childbearing potential must agree to use a highly effective method of contraception throughout the study and for a minimum of 90 days after the last dose of treatment on protocol. A patient is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active. Female patients who are not of childbearing potential should meet at least one of the following criteria:

  * Have undergone hysterectomy or bilateral oophorectomy; or
  * Have medically confirmed ovarian failure; or
  * Are medically confirmed to be post-menopausal (cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause

Exclusion Criteria:

* Lymphoblastic crisis of CML
* Mature B cell (Burkitt's) ALL
* Active central nervous system (CNS) leukemia, as defined by unequivocal morphologic evidence of lymphoblasts in the cerebrospinal fluid (CSF), use of CNS-directed local treatment for active disease within the prior 28 days, symptomatic CNS leukemia (i.e., cranial nerve palsies or other significant neurologic dysfunction) within 28 days. Prophylactic intrathecal medication is not a reason for exclusion.
* Pregnant women or women who are breast-feeding
* Concurrent active malignancy requiring immediate therapy
* Patients with human immunodeficiency virus (HIV)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
proportion of patients who have a dose limiting toxicity (DLT) | with in 6 weeks of starting the study drug
  DLTs are defined as any of the following: grade 4 pancreatitis, grade 4 hemorrhage, grade 4 thromboembolism, grade 4 hyperbilirubinemia and any grade 5 toxicity attributable (definitely, probably or possible) to Erwinia asparaginase.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/